CLINICAL TRIAL: NCT03660410
Title: Study of Oral Conditions in Indigenous Populations in the State of Roraima - Brazil
Status: Completed | Type: Observational
Sponsor: Universidade Metropolitana de Santos (Other)
Responsible Party: Principal Investigator, CAIO VINICIUS GONÇALVES ROMAN TORRES, Professor Doctor, Universidade Metropolitana de Santos
Other Study IDs: SantosMU03
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Diagnosis, Oral; Periodontal Diseases; Caries, Dental
Keywords: indians, south american; periodontal disease; dental caries
MeSH Terms: conditions — Disease; Periodontal Diseases; Dental Caries | interventions — Immunologic Memory; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Yanomamis: Yanomami Indians, Anamnesis and oral clinical examination
  Interventions: Other: Anamnesis; Other: Oral clinical examination
- Macuxi: Macuxi Indians, Anamnesis and oral clinical examination
  Interventions: Other: Anamnesis; Other: Oral clinical examination
- Wapixana: Wapixana Indians, Anamnesis and oral clinical examination
  Interventions: Other: Anamnesis; Other: Oral clinical examination

INTERVENTIONS:
Other: Anamnesis — A detailed anamnesis should be carried out in order to know the habits, the presence of systemic pathologies, the use of medication
Other: Oral clinical examination — Clinical examination should be carried out evaluating the presence of caries, tooth loss, periodontal condition, occlusal factors

SUMMARY:
The objective of this cross - sectional observational study will be to evaluate the oral conditions of indigenous people in the state of Roraima, comparing habits and hygiene conditions in each ethnicity evaluated. This project was submitted to the Coordination of the Yanomami Indigenous Special Sanitary District, the CONDISI presidency and the CASAI leadership. Around 200 indigenous people from the aforementioned ethnic groups, of both sexes, aged between 18 and 75 years, will be evaluated

DETAILED DESCRIPTION:
The indigenous population, as well as the non-indigenous population, has been plagued by oral diseases throughout its history. Within the population in general, periodontal diseases exhibit great expressiveness, they appear as the most common chronic diseases, but in the indigenous population there is a certain epidemiological invisibility. In this population there is a shortage in the studies, some of these show that the higher prevalences of insertion level and depth of probing occur in individuals with more advanced age and that they are afflicted with periodontal diseases. The objective of this cross - sectional observational study will be to evaluate the oral conditions of indigenous people in the state of Roraima, comparing habits and hygiene conditions in each ethnicity evaluated. This project was submitted to the Coordination of the Yanomami Indigenous Special Sanitary District, the CONDISI presidency and the CASAI leadership. Around 200 indigenous people from the aforementioned ethnic groups, of both sexes, aged between 18 and 75 years, will be evaluated, with voluntary participation and by means of the signature of the free and informed consent form of the same or its person in charge. Due to the difficulties encountered in the indigenous communities in relation to the distance from health care, where there are no care centers near their residence and thus not obtaining the information necessary for basic health care, with the aggravation of contact with the culture. Indigenous people with often deleterious eating habits, we expect to find a population with many oral health problems, such as periodontal disease, dental caries and tooth loss. The insufficiency of studies with appropriate methodology gives the indigenous peoples of Latin America an epidemiological invisibility that impairs the production of knowledge about oral health conditions and the elaboration of strategies to prevent oral diseases and promote health in these populations.

ELIGIBILITY:
Inclusion Criteria:

* individuals of the Macuxi, Yanomami and Wapixana ethnic groups aged between 18 and 75 years

Exclusion Criteria:

* Individuals who have included periodontal treatment in the last 6 months;
* hospitalized with antibiotic therapy in the last 6 months;
* who need medication for clinical evaluation and
* total edentulous individuals.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the present study, about 200 indigenous people of the Yanomami, Macuxi and Wapixana ethnic groups of both genders, aged between 18 and 75 years, were evaluated in their respective communities located in the state of Roraima.
  Clinical parameters evaluated were Depth of Depth (PS), Clinical Insertion Level (NCI), Index of Plaque (PI), Bleeding Index (IS), Caries Index, Lost and Sealed Index (DMFT); The examiners were previously calibrated by means of periodontal clinical parameters measurements and compared intra-examiner and inter-examiner. Data were tabulated and received adequate statistical treatment (p <0.05).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Probing Deep | 1 day
  probing deep in six points/teeth

SECONDARY OUTCOMES:
Gingival index | 1 day
  gingival index in four points / teeth
Plaque index | 1 day
  plaque index in four points/teeth

CONTACTS AND LOCATIONS:
Locations (1):
- Caio Vinicius Gonçalves Roman Torres, Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No